CLINICAL TRIAL: NCT05141058
Title: T Cell Therapy Opposing Novel COVID-19 Infection in Immunocompromised Patients
Acronym: TONI
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Susan Conway, Critical Medicine Physician, Children's National Research Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: TONI
Record Dates: First submitted 2021-11-10; First posted 2021-12-02 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Adults (18 to <80 years) (Experimental): Arm A will include adult participants who are at least 18 years of age but younger than 80 years.
  Interventions: Biological: Coronavirus-specific T cell (CST)
- Older children (12 to <18 years) (Experimental): Arm B will include adolescent participants who are at least 12 years of age but younger than 18 years.
  Interventions: Biological: Coronavirus-specific T cell (CST)
- Young children (2 to <12 years) (Experimental): Arm C will include pediatric participants who are at least 2 years of age but younger than 12 years.
  Interventions: Biological: Coronavirus-specific T cell (CST)

INTERVENTIONS:
Biological: Coronavirus-specific T cell (CST) — Participants will receive donor-derived CSTs for prevention of SARS-CoV-2 infection after HSCT (≥28 days and <4 months after hematopoietic stem cell transplantation (HSCT).

SUMMARY:
This is an open label, phase I dose-escalation study to evaluate the safety of coronavirus-specific T cell (CST) therapy for prevention of SARS-CoV-2 infection in immunocompromised patients following hematopoietic stem cell transplantation (HSCT).

Participants will receive donor-derived CSTs for prevention of SARS-CoV-2 infection after HSCT (≥28 days and <4 months after HSCT).

In this dose escalation trial, three doses (1x107/m2, 2x107/m2, and 4x107/m2) will be tested for safety, with study arms for adult (≥18 years of age and <80 years) HSCT recipients (Arm A) and two arms for pediatric (≥12 years of age and <18 years; ≥2 years and <12 years) HSCT recipients (Arm B and Arm C, respectively), and defined dose escalations in each study arm. The study agent will be assessed for safety (stopping rules defined) and antiviral activity.

DETAILED DESCRIPTION:
The primary purpose of this phase I study is to assess the safety of administering donor-derived CSTs in immunocompromised participants for prevention of SARS-CoV-2 infection. Related and unrelated donors of participants who are at risk of SARS-CoV-2 infection will be enrolled for screening and production of CSTs from peripheral blood. Following product manufacturing, participants who have undergone HSCT will receive donor-derived CSTs for prevention of SARS-CoV-2 infection.

It is a dose escalation study with separate study arms for adult (Arm A) and pediatric (Arms B and C) recipients of HSCT who are at risk of SARS-CoV-2 infection. Participants who have undergone HSCT and test negative for SARS-CoV-2 infection will be enrolled and receive one dose of CST product derived from their HSCT donor for prophylaxis. Participants aged ≥18 years and <80 years will be enrolled on Arm A, participants who are ≥12 years of age and <18 years of age will be enrolled on Arm B, and participants who are ≥2 years of age and <12 years of age will be enrolled on Arm C.

Investigators will test three doses: 1x107 /m2, 2x107 /m2, and 4x107 /m2. At least 3 adult participants (Arm A) will be enrolled at each dose level before pediatric participants (Arm B) are enrolled. At each dose level, treatment of the first two adult participants enrolled at that dose level will be staggered at least 28 days apart and each will be followed for the 45-day safety monitoring period to assess safety and efficacy of CST product. Once the third adult participant on any given dose level has completed their 45-day safety monitoring period and the safety and efficacy data is reviewed and approved by the FDA, then adult participants can be escalated to the next dose level and pediatric participants can start enrollment at the dose level completed by the adult participants. If participants show evidence of safety and at least 2 of 3 have evidence of antiviral immune reconstitution against SARS-CoV-2, investigators will enroll pediatric participants at that dose level following FDA approval.

Additionally, infusion of pediatric participants enrolled at each dose level will be staggered at least 28 days apart, and all enrolled participants will be followed for 45 days for safety monitoring after CST infusion.

After receiving the CST infusion, participants will be closely monitored to evaluate their health status and the effects of treatment. Follow-up visits will occur frequently and will continue for up to 1 year after the CST infusion. During these visits, study doctors will perform clinical assessments, including medical history and physical examinations. Blood tests will be conducted, such as complete blood count (CBC) and comprehensive metabolic panel (CMP), and research blood samples will also be collected for analysis. These assessments will help monitor safety, toxicity, and treatment effects.

ELIGIBILITY:
Inclusion Criteria:

Participant Inclusion Criteria for CST Infusion:

1. For recipient of CSTs derived from an HSCT donor under Arm A:

   a. Patients aged ≥18 years and <80 years who were recipients of prior myeloablative or non-myeloablative allogeneic HSCT using either bone marrow or peripheral blood stem cells or single or double cord blood ≥28 days and <4 months ago who are at risk of SARS-CoV-2 infection.
2. For recipient of CSTs derived from an HSCT donor under Arms B and C:

   a. Patients aged ≥2 years and <18 years who were recipients of prior myeloablative or non-myeloablative allogeneic HSCT using either bone marrow or peripheral blood stem cells or single or double cord blood ≥28 days and <4 months ago who are at risk of SARS-CoV-2 infection.
3. Have evidence of primary engraftment following HSCT (defined by ANC ≥500/mm3 for three consecutive measurements on different days, respectively)
4. Participants receiving calcineurin inhibitors for treatment of GVHD, or for other reasons, should not have any dosage changes within 7 days prior to infusion**

   a. For patients receiving steroids, dosage must have been tapered to <0.5 mg/kg/day of prednisone (or equivalent) at least 7 days prior to infusion.
5. Karnofsky/Lansky score >70.
6. ≥2 years to <80 years of age at enrollment.
7. Absolute neutrophil count (ANC) ≥500/ul.
8. Hemoglobin ≥8.0g/dl (level can be achieved with transfusion).
9. Platelets ≥20 K/ul (level can be achieved with transfusion)*.
10. Bilirubin ≤2x upper limit normal.
11. Aspartate transaminase (AST) ≤2.5x upper limit of normal.
12. Alanine transaminase (ALT) ≤2.5x upper limit of normal.
13. Estimated GFR >60mL/min/1.73m2 (calculated per institutional standards).
14. Pulse oximetry of ≥92% on room air for at least 7 days prior to infusion.
15. Age appropriate mean arterial pressure without the use of vasopressors.
16. Negative pregnancy test in female participant of childbearing potential.
17. Male and female participants of childbearing potential must use highly effective birth control measures or practice abstinence for a minimum of 6 months after receiving study therapy
18. Written informed consent and/or signed assent line from participant, parent or guardian.

Donor Inclusion Criteria:

1. Donors for allogeneic (i.e. HLA matched or mismatched related or unrelated) stem cell transplants who have fulfilled eligibility as per FDA regulations outlined in 21 Code of Federal Regulations (CFR) 1271 subpart C. This includes that donors have been deemed in good health by donor physician based on physical examination and laboratory testing. If a donor has been chosen for the transplant based on urgent medical need that same donor will also be used for CST generation provided that there are no new reasons for ineligibility since the stem cell collection.
2. Donor or guardian of pediatric donor capable of providing informed consent.
3. 2 to 80 years of age.
4. Female donors of childbearing potential must have a negative pregnancy test.

Exclusion Criteria:

Participants Exclusion Criteria for CST Infusion:

1. Participants receiving biological or immunosuppressive monoclonal antibodies targeting T cells within 28 days prior to CST infusion, including ATG, Alemtuzumab, Basiliximab, Tociluzimab, Brentuximab, or other medications under this category as determined by the investigators.

   a. If alemtuzumab has been received within 6 weeks prior to CST infusion, plasma levels should be obtained to ensure drug clearance (≤0.16 pg/ml).
2. Participants who have received donor lymphocyte infusion (DLI), chimeric antigen receptor T cell infusion, or other experimental cellular therapies within 28 days prior to CST infusion.
3. Participants who have received ruxolitinib or other JAK inhibitors within 7 days prior to CST infusion.
4. Participants with uncontrolled or progressing infections or active infections causing fever (temperature ≥38.1°C). Uncontrolled infections are defined as bacterial, fungal, or viral infections (including HIV and Hepatitis B and C) with either clinical signs of worsening despite standard therapy that may be attributed to the uncontrolled infection. Progressing infection is defined as hemodynamic instability, worsening physical signs, or radiographic findings attributable to infection.

   1. For bacterial infections, participants must be receiving definitive therapy and have no signs of progressing infection within 7 days prior to CST infusion.
   2. For fungal infections, participants must be receiving definitive systemic anti-fungal therapy and have no signs of progressing infection within 7 days prior to CST infusion.
5. Participants with unexplained fever (temperature ≥38.1°C) within 7 days prior to CST infusion.
6. Participants with evidence of active SARS-CoV-2 infection based on SARS-CoV-2 RT-PCR positivity.
7. Participants with hypotension (mean arterial pressure <50mmHg in participants <5 years of age, <55 mmHg in participants ≥5 and <14 years of age or <60 mmHg in participants ≥14 years of age).
8. Participants with pulse pressure >40 mmHg.
9. Participants with respiratory rate >20 breaths per minute.
10. Participants with heart rate ≥140 beats per minute.
11. Participants with uncontrolled hypertension as defined by systolic blood pressure >99th percentile for age (participants <18 years), and systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg (participants ≥18 years).
12. Participants with metabolic instability.
13. Pediatric participants with modified Ross heart failure Class II disease and adult participants with NYHA Class II disease.
14. Participants with advanced pulmonary disease as defined by requirement for supplemental oxygen or positive pressure ventilation due to pulmonary disease. (This includes participants with active interstitial lung disease (ILD)/pneumonitis, advanced pulmonary disease, a history of ILD/pneumonitis requiring treatment with systemic steroids or a baseline oxygen requirement).
15. Participants with neurological or psychiatric disorders that would, in the opinion of the investigators, place them at increased risk of harm, impact the investigator's abilities to screen for adverse events in the subject, or impair the subject's ability to provide informed consent.
16. Participants receiving checkpoint inhibitors within the previous 3 months prior to CST infusion, including nivolumimab, pembroluzimab, or other related medications.
17. Participants with proven or suspected MIS (in both adults and children) based on the CDC definition and investigator judgement.
18. Participants who are breastfeeding.
19. Participants who have received live vaccines within 30 days, or any SARS-CoV-2 vaccine in the past 28 days prior to enrollment.
20. Participants with any other unrelated medical conditions that would impact the participant's safety in the opinions of the investigators.
21. Participants anticipated to need a blood transfusion within 48 hours of CST infusion.
22. Participants unwilling to utilize effective contraception during the study period (if applicable)

Donor Exclusion Criteria:

1. Donation of cells would pose a physical or psychological risk to the donor.
2. Prior or current complicated course of COVID-19, including but not limited to MIS, CRS, or thromboembolic complications based on investigator judgement.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-10-19 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade ≥3 infusion-related Adverse Events (AEs) | Within 45 days of CST infusion
  Number of patients with grade ≥3 infusion-related AEs at 45 days of following CST infusion.
Incidence of acute Graft Vs Host Disease (aGVHD) grade ≥3 | Within 45 days of CST infusion
  Number of patients with aGVHD grade ≥3 within 45 days of CST infusion.
Incidence of Systemic Inflammatory Response Syndrome (SIRS) or CRS | Within 45 days of CST infusion
  Number of patients with systemic Inflammatory Response Syndrome (SIRS) or CRS
Incidence of Multi-System Inflammatory Syndrome (MIS) | Within 45 days of CST infusion
  Number of patients with MIS

SECONDARY OUTCOMES:
COVID-19 antiviral immunity using intracellular flow cytometry | At 45 days following CST infusion
  Participant serum and PBMCs will be monitored for COVID-19 virus specific T cell activity at 45 days following CST infusion by phenotypic and functional studies including ELIspot with appropriate viral specific peptide mixtures and available HLA-restricted epitope peptides, intracellular cytokine staining, serum cytokine profiling and/or other assays as they become available for immune profiling purposes
COVID-19 antiviral immunity using intracellular ELIspot assays | At 45 days following CST infusion
  Participant serum and PBMCs will be monitored for COVID-19 virus specific T cell activity at 45 days following CST infusion by phenotypic and functional studies including ELIspot with appropriate viral specific peptide mixtures and available HLA-restricted epitope peptides, intracellular cytokine staining, serum cytokine profiling and/or other assays as they become available for immune profiling purposes
Persistence of infused CSTs | Within 12 months
  Persistence of infused T cells will be monitored using deep sequencing to track the TCRB repertoire in the participant peripheral blood
Antiviral Activity | Within 12 months
  Antiviral activity will be assessed by measurement of SARS-CoV-2 viral load by screening RT-PCR from oral/salivary samples or from respiratory samples for any participant who develops a positive SARS-CoV-2 RT-PCR post CST infusion

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Children's National Hospital, Washington D.C., District of Columbia
  - The Sidney Kimmel Comprehensive Cancer Center, Johns Hopkins University, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No